CLINICAL TRIAL: NCT05208359
Title: Supporting Refugee and Immigrant Youth's Mental Health: Examining Effectiveness and Implementation of a School-Based Intervention
Brief Title: Supporting Refugee and Immigrant Youth's Mental Health
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Loyola University Chicago (Other)
Collaborators: Ann & Robert H Lurie Children's Hospital of Chicago (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2783; R15MH128722 (NIH)
Record Dates: First submitted 2021-12-14; First posted 2022-01-26 (Actual); Results first posted 2025-07-11 (Actual); Last update posted 2025-07-11 (Actual); Status verified 2025-06

CONDITIONS: Mental Health
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- STRONG immediate group (Experimental): Small mental health support group delivered immediately
  Interventions: Behavioral: Supporting Transition Resilience Of Newcomer Groups (STRONG)
- STRONG delayed group (Other): Small mental health support group delivered after a delay of approximately 3 months
  Interventions: Behavioral: Supporting Transition Resilience Of Newcomer Groups (STRONG)

INTERVENTIONS:
Behavioral: Supporting Transition Resilience Of Newcomer Groups (STRONG) — 10 group sessions that offer skills, strengths, support, and affirmation for newcomer youth

SUMMARY:
The purpose of this study is to examine the effectiveness of STRONG on the mental health of refugee and immigrant students using a group randomized waitlist control design (e.g., randomization by school/group). Further, the impact of STRONG on key target mechanisms (e.g., resilience, coping, and school connectedness) are also examined. Finally, investigators examine the implementation of STRONG to guide additional dissemination. School-based mental health clinicians will co-facilitate STRONG groups in schools, meeting once a week. STRONG will be implemented in six public schools across two academic years. In each school, one group of approximately five students will be implemented, resulting in a sample of 60 students total across the two years. Schools will be randomly assigned to either provide the STRONG program immediately (immediate treatment) or after three months (delayed treatment). A team of 10 undergraduate students and four graduate students will collect data at baseline and at three- and six-months post baseline.

Aim 1: Evaluate impact of STRONG on student mental health via randomized waitlist control design.

1) Investigators hypothesize that students who participate in STRONG will show improvements in self-reported, parent-reported, and teacher-reported mental health (emotional symptoms, conduct problems, hyperactivity/inattention, and peer problems) as compared to the waitlist control group (primary outcome).

Aim 2: Examine the impact of STRONG on resilience, coping, and school connectedness and how these changes are related to student mental health outcomes.

1. Investigators hypothesize that students who participate in STRONG will show improvements in self-reported resilience, coping efficacy, school connectedness, and parent-reported coping as compared to the waitlist control group (target mechanisms).
2. Investigators hypothesize that these changes will be related to student mental health improvement/maintenance over time (mechanism of action).

Aim 3: Examine implementation of STRONG across schools.

1. Investigators will conduct focus groups with clinicians and interviews with school personnel (teachers, administrators) to examine the challenges and successes related to implementation of STRONG. Qualitative thematic analysis will be conducted.
2. Satisfaction (clinician, parent, and student), student engagement with each session, and fidelity ratings will be examined.

DETAILED DESCRIPTION:
STRONG will be implemented in six public schools during 2021-2022 academic year and six public schools during the 2022-2023 academic year. Investigators anticipate three elementary schools and three high schools each year. Within CPS, school leadership has requested interventions specifically designed for refugee and immigrant students due to school population and need. In each school, one group of approximately five students will be implemented. Schools will be randomly assigned to either provide the STRONG program immediately (immediate treatment) or after three months (delayed treatment). Randomization will include balancing of elementary and high schools so that the number of elementary and high schools randomized to immediate vs. delayed treatment will be equivalent. School mental health staff (e.g., district-employed social workers or community clinicians who provide services in schools) will co-facilitate groups in schools, meeting once a week. School-based clinicians are typically expected to deliver one to two small group interventions as part of their job duties. District partners have committed to supporting clinicians in delivering STRONG as part of this expectation. The research team, comprised of 10 undergraduate students and four graduate students, will collect data at baseline and then at three- and six-months post baseline. Undergraduate and graduate student pairs will meet with students and parents at schools allowing for support and mentorship of undergraduate research assistants along with clinical expertise from graduate students enrolled in the Clinical Psychology PhD program at Loyola University Chicago.

Eligibility Criteria Students will be identified by trained STRONG clinicians consistent with standard school procedures, which include teacher and other school staff referral, parent nomination, and clinician identification from other support services. Eligibility criteria include (1) newcomer status (students who have migrated to a new country) and (2) difficulties in functioning or coping as assessed by school staff (teacher, school-based clinician). Referral reasons may include general difficulties, academic performance, peer relationships, family relationships, physical problems, behavioral concerns, and/or appearance of affect, among others. The eligibility criteria are intentionally designed to be broad (i.e., not a strict clinical cutoff) with the purpose of being more inclusive, understanding that cultural and environmental differences may produce different behavioral and emotional outcomes than what typical clinical assessments capture. In addition, researchers call for mental health treatment for refugee and immigrant children that can address trauma, acculturation, isolation, and resettlement, to better address needs. Due to the diversity in experiences, this can also impact the presenting concerns of children during the resettlement process. Thus, it is important to have a broader inclusion criterion to best fit the needs of this group. This way children that may not be presenting with solely PTSD symptoms, including anxiety, depression, and stress management problems can also benefit from a mental health intervention that highlights their strengths. STRONG allows for this flexibility needed in addressing presenting concerns among this diverse population.

Intervention Training for clinicians to implement STRONG will occur in fall 2021. Training will be facilitated by the Center for Childhood Resilience (CCR) at Lurie Children's Hospital. The STRONG training is two days and provides an overview of each session, practice of strategies, and implementation planning. STRONG includes 10 small group sessions, one individual session (for journey narrative), and teacher and parent education sessions. There is an elementary and high school version of the manual, modified for developmental appropriateness (Hoover et al., 2019). Group sessions include recognizing internal strengths, identifying family/social supports, relaxation, mindfulness, cognitive coping, and problem-solving. Each session includes newcomer-specific examples and support for students in applying strategies to their newcomer experience as well as natural opportunities to foster positive identity and build on strengths.

In the elementary and high school groups, session one helps students identify internal strengths and external support systems (family/social supports), while in session two students learn about stress and how it impacts their bodies and minds. In the third session, stress reactions and feeling identifications are explored, and in the fourth session feelings management is discussed. In session five, students begin the session by sharing an object that represents where they are from, fostering positive cultural identity. Then, students begin to explore the cognitive aspect of mental health and learn about using helpful thoughts. In session six, children learn about the "steps to success", in which they create goals and manageable steps to achieve them, as well as ways to address avoidance. In session seven, children are taught different strategies for problem solving. In session eight, students share something meaningful from their home country (e.g., favorite food, special place, favorite tradition) and then share parts of their journey with the group. In the ninth session, students share about a favorite holiday or tradition and then continue sharing about their journeys. Then in session 10, students take turns appreciating strengths they have noticed about group members and then take part in a graduation celebration. Between sessions four and eight, students meet individually with the clinician to discuss their journey to the U.S. This may include positive and difficult experiences, including potential traumatic experience. The clinician guides students to recognize strengths that helped them get through their journey rather than focusing on a single event with repeated retelling. The journey narrative is flexible to allow students to discuss multiple traumatic experiences, while also highlighting strengths and assets. It is recommended that the clinician screen for significant PTSD symptoms in individual sessions to consider if additional referrals will be necessary after STRONG. Clinicians also have individual sessions with caregivers and teachers to provide psychoeducation on the children's participation in the STRONG program. This allows for caregivers and teachers to support the student's progress in multiple settings.

Participants An estimated 60 students will participate in STRONG (five students per group across six public schools over two years). Student age range will be 8-18, though each STRONG group will be comprised of students within one grade level of each other. Clinicians, school personnel (teachers, administrators), and parents will be invited to complete measures and participate in focus groups (clinicians) or interviews (teachers, administrators). Teachers who have students participating in STRONG and/or assisted with referrals/identification of students will be recruited to participate in interviews. Teacher participants will be identified in collaboration with school partners/administrators. For example, English Language Learner (ELL) teachers have been key partners in referrals/identification of students in our preliminary feasibility pilot.

Procedure Clinicians will identify eligible students and reach out to parents/caregivers consistent with standard school procedures. Clinicians will offer a group or individual information meeting to share more about STRONG and will ask parent permission to share contact information with the research team. With permission, the research team will meet with parents as part of the informational meeting or at a later date to provide additional information about the research protocol and obtain informed consent and assent.

Data will be collected from students, parents, and teachers at baseline and then at three- and six-months post baseline. Questionnaires will include measures of emotional/behavioral symptoms as well as coping and resilience. Caregivers will also be asked to provide demographic information. The three-month assessment point will represent "post-intervention" data for students at schools randomized to immediate treatment, and will be a second "pre-intervention" time-point for students at schools randomized to delayed treatment. The six-month assessment will represent three-month follow-up data for students at schools randomized to immediate treatment and "post- intervention" data for students at schools randomized to delayed treatment. School-based mental health staff will complete fidelity monitoring forms after each session, and will provide quantitative and qualitative feedback on their satisfaction with the program.

ELIGIBILITY:
Inclusion Criteria:

* newcomer status (students who have migrated to a new country)
* difficulties in functioning or coping as assessed by school staff (teacher, school-based clinician).

Exclusion Criteria:

* Born in mainland United States

Ages: 8 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 64 (Actual)
Dates: Start 2021-11-04 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-07-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Loyola University Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Yes
Data have been deposited into NIMH Data Archive.
Time Frame: The data has been deposited in NIMH Data Archive.
Access Criteria: Accessible via NIMH Data Archive

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible newcomer students were identified by school staff (teachers, school-based clinicians) across 6 participating schools.
Pre-assignment Details: Of the 84 identified students, 64 students were assigned to treatment groups. Students not assigned to either treatment groups declined consent, moved schools, or could not be reached.
Units Other Than Participants: groups
Period: Overall Study
Arm/Group | STRONG Immediate Group | STRONG Delayed Group
Started | 32; 6 groups | 32; 6 groups
Completed | 32; 6 groups | 32; 6 groups
Not Completed | 0; 0 groups | 0; 0 groups

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | STRONG Immediate Group | STRONG Delayed Group | Total
Number analyzed (Participants) | 32 | 32 | 64
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.13 (3.17) | 14.66 (2.90) | 13.89 (3.11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 8 | 29
  Male | 11 | 24 | 35
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African American/Black | 3 | 2 | 5
  Asian | 8 | 14 | 22
  Latiné/Hispanic | 16 | 12 | 28
  MENA | 5 | 3 | 8
  Missing | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 32 | 32 | 64
Strengths and Difficulties Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Stress and Difficulties Questionnaire (SDQ) is a 25-item (e.g., "I worry a lot") questionnaire with four subscales: emotional symptoms, conduct problems, hyperactivity/inattention problems, and peer problems. Participants answer on a 3-point Likert scale (0 = "Not at All" to 2 = "Certainly True"). Externalizing Problems are the sum of the conduct problems and hyperactivity scales. Internalizing Problems are the sum of emotional symptoms and peer problems. Scales mean range from 0 to 20 total points, with higher scores reflecting higher problems.
  units on a scale
    Internalizing Problems (self-report) | 4.70 (2.73) | 3.71 (2.92) | 4.20 (2.85)
    Internalizing Problems (teacher-report) | 2.46 (2.08) | 1.84 (1.65) | 2.15 (1.89)
    Externalizing Problems (self-report) | 6.34 (4.02) | 5.40 (3.13) | 5.87 (3.60)
    Externalizing Problems (teacher-report) | 4.27 (4.07) | 4.58 (4.21) | 4.43 (4.11)
Connor-Davidson Resilience Scale [Mean (Standard Deviation); unit: units on a scale] — Connor-Davidson Resilience Scale is a 25-item measures that measures adaptability and resilience among youth. Participants rated each item on a 5-point Likert scale (0= "Not True at All" to 4 = "True Nearly All of Time"). Total scores range from 0 to 100, with higher scores indicating more adaptability and resilience.
  units on a scale | 69.62 (12.03) | 67.24 (16.02) | 68.43 (14.11)
The Coping Efficacy Scale [Mean (Standard Deviation); unit: units on a scale] — The Coping Efficacy Scale (Sandler et al., 2000) measures an individual's belief in their ability to use coping strategies to handle future stressors and novel situations. For this study, six items designed to assess both satisfaction with past coping efforts and anticipated effectiveness in handling future problems were included. The scale uses a 4-point scale (1= "Not At All" to 4 = "Well") where higher scores indicate greater coping efficacy. Mean scores were used.
  units on a scale
    Self-report | 3.12 (0.51) | 2.96 (0.67) | 3.04 (0.60)
    Caregiver-report | 3.21 (0.77) | 3.13 (0.67) | 3.17 (0.71)
Responses to Stress Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Responses to Stress Questionnaire (RSQ) is a 57-item multidimensional measure on 4-point Likert scale (1= "Not at all" to 4 = "A lot"). Primary control, secondary control, and disengagement coping factors were used in this study. With higher mean scores reporting higher coping in each respective factor.
  units on a scale
    Primary control coping | 2.50 (0.47) | 2.46 (0.68) | 2.48 (0.58)
    Secondary control coping | 2.66 (0.63) | 2.63 (0.55) | 2.65 (0.59)
    Disengagement coping | 2.14 (0.74) | 2.22 (0.66) | 2.18 (0.70)
School Connectedness Scale [Mean (Standard Deviation); unit: units on a scale] — The School Connectedness Scale is a 5-item questionnaire that measures youth's bond toward their school on a 5-point Likert scale (1="Strong Disagree" to 5="Strongly Agree"). Mean scores were used in analysis, with higher scores indicating higher school connectedness.
  units on a scale | 4.26 (0.81) | 4.07 (0.75) | 4.16 (0.78)

OUTCOME MEASURES:

1. Primary Outcome: Strengths and Difficulties Questionnaire
Description: The Stress and Difficulties Questionnaire is a 25-item (e.g., "I worry a lot") questionnaire with four subscales: emotional symptoms, conduct problems, hyperactivity/inattention problems, and peer problems. Participants answer on a 3-point Likert scale (0 = "Not at All" to 2 = "Certainly True"). Externalizing Problems are the sum of the conduct problems and hyperactivity scales. Internalizing Problems are the sum of emotional symptoms and peer problems. Scales mean range from 0 to 20 total points, with higher scores reflecting more problems (e.g., worse outcome).
Time Frame: Baseline, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STRONG Immediate Group | STRONG Delayed Group
Number analyzed (Participants) | 32 | 32
units on a scale
  Self-reported internalizing (3 months) | 4.91 (2.42) | 3.49 (2.49)
  Teacher-reported internalizing (3 months) | 2.72 (2.71) | 2.72 (2.53)
  Self-reported internalizing (6 months) | 4.05 (2.26) | 3.09 (2.23)
  Teacher-reported internalizing (6 months) | 2.40 (2.50) | 2.40 (2.06)
  Self-reported externalizing (3 months) | 5.85 (3.71) | 6.20 (3.24)
  Teacher-reported externalizing (3 months) | 3.75 (4.31) | 5.65 (4.50)
  Self-reported externalizing (6 months) | 5.40 (3.53) | 5.07 (2.90)
  Teacher-reported externalizing (6 months) | 4.23 (4.45) | 5.41 (3.53)

2. Secondary Outcome: Connor-Davidson Resilience Scale
Description: Connor-Davidson Resilience Scale is a 25-item measures that measures adaptability and resilience among youth. Participants rated each item on a 5-point Likert scale (0= "Not True at All" to 4 = "True Nearly All of Time"). Total scores range from 0 to 100, with higher scores indicating more adaptability and resilience (e.g., better outcome).
Time Frame: Baseline, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STRONG Immediate Group | STRONG Delayed Group
Number analyzed (Participants) | 32 | 32
units on a scale
  3 months | 75.68 (16.46) | 72.08 (14.54)
  6 months | 74 (15.15) | 75.27 (11.65)

3. Secondary Outcome: The Coping Efficacy Scale
Description: The Coping Efficacy Scale (Sandler et al., 2000) measures an individual's belief in their ability to use coping strategies to handle future stressors and novel situations. For this study, six items designed to assess both satisfaction with past coping efforts and anticipated effectiveness in handling future problems were included. The scale uses a 4-point scale (1= "Not At All" to 4 = "Well"), with higher scores indicating greater coping efficacy (e.g., better outcome).
Time Frame: Baseline, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STRONG Immediate Group | STRONG Delayed Group
Number analyzed (Participants) | 32 | 32
units on a scale
  Self-reported (3 months) | 2.98 (0.55) | 3.09 (0.53)
  Caregiver-reported (3 months) | 3.30 (0.51) | 3.14 (0.82)
  Self-reported (6 months) | 3.05 (0.58) | 3.10 (0.60)
  Caregiver-reported (6 months) | 3.44 (0.55) | 3.12 (0.81)

4. Secondary Outcome: Responses to Stress Questionnaire
Description: The Responses to Stress Questionnaire (RSQ) is a 57-item multidimensional measure on 4-point Likert scale (1= "Not at all" to 4 = "A lot"). Primary control, secondary control, and disengagement coping factors were used in this study. With higher mean scores reporting higher coping in each respective factor. Mean scores were used.
Time Frame: Baseline, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STRONG Immediate Group | STRONG Delayed Group
Number analyzed (Participants) | 32 | 32
units on a scale
  Primary coping (3 months) | 2.63 (0.67) | 2.47 (0.62)
  Secondary coping (3 months) | 2.70 (0.46) | 2.67 (0.63)
  Disengagement coping (3 months) | 2.08 (0.67) | 2.08 (0.67)
  Primary coping (6 months) | 2.82 (0.57) | 2.60 (0.66)
  Secondary coping (6 months) | 2.66 (0.52) | 2.62 (0.55)
  Disengagement coping (6 months) | 2.01 (0.64) | 2.09 (0.75)

5. Secondary Outcome: School Connectedness Scale
Description: The School Connectedness Scale is a 5-item questionnaire that measures youth's bond toward their school on a 5-point Likert scale (1="Strong Disagree" to 5="Strongly Agree"). Mean scores were used in analysis, with higher scores indicating higher school connectedness (e.g., better outcome).
Time Frame: Baseline, 3 months, and 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | STRONG Immediate Group | STRONG Delayed Group
Number analyzed (Participants) | 32 | 32
units on a scale
  3 months | 4.27 (0.52) | 4.11 (0.78)
  6 months | 4.17 (0.75) | 4.08 (0.86)

ADVERSE EVENTS:
Time Frame: 1 year, 7 months
Description: 0 participants experiences all-cause mortality and serious adverse events. 1 participant experienced 1 other (not including serious) adverse event through self-disclosure from participant to research assistant during data collection.
Arm/Group | STRONG Immediate Group | STRONG Delayed Group
All-Cause Mortality (participants affected / at risk) | 0/32 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/32 | 0/32
Other Adverse Events (participants affected / at risk) | 0/32 | 1/32
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | STRONG Immediate Group (N=32) | STRONG Delayed Group (N=32)
Endorsed risk and abuse (Social circumstances) | 0 (0) | 1 (1) — Passive suicidal ideation was endorsed and risk assessment was conducted. Potential verbal and physical abuse were reported to the Department of Child and Family Services.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Addition of Cover Page (2025-02-14): https://cdn.clinicaltrials.gov/large-docs/59/NCT05208359/Prot_SAP_002.pdf
  • Informed Consent Form: Parent Consent English (2022-07-13): https://cdn.clinicaltrials.gov/large-docs/59/NCT05208359/ICF_003.pdf
  • Informed Consent Form: Child Assent English (2021-10-19): https://cdn.clinicaltrials.gov/large-docs/59/NCT05208359/ICF_004.pdf